CLINICAL TRIAL: NCT01028599
Title: Effect of Physical Training on Oxygen Uptake and Endothelial Function in Heart Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, Dr, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-D-2009-004
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Transplantation; Exercise Capacity; Endothelial Function
Keywords: Heart transplantation; Exercise capacity; Endothelial function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Other: Intensive physical exercise

INTERVENTIONS:
Other: Intensive physical exercise — Intensive physical exercise 1 hour three times per week

SUMMARY:
The purpose of this study is to investigate the effect of physical training on work capacity and vascular function after heart transplantation, cardiac transplant recipients are randomized to 8 weeks of intense physical training or control. Vascular function is measured non-invasively. Effect on the hormones and the immune system is evaluated using blood samples.

DETAILED DESCRIPTION:
To investigate the effect of physical training on work capacity and vascular function after heart transplantation, cardiac transplant recipients are randomized to 8 weeks of intense physical training or control. Vascular function is measured non-invasively using forearm flow mediated dilatation. Effect on the blood natriuretic peptides and the inflammatory markers is evaluated using blood samples at baseline and after the training or control period.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant recipients > 1 year after transplantation

Exclusion Criteria:

* Recent rejection, severe renal dysfunction, graft dysfunction, allograft vasculopathy, cancer, inability to exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in maximal oxygen uptake. | 8 weeks

SECONDARY OUTCOMES:
Change inm flow mediated vasodilatation. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, PhD, Principal Investigator — Department of Cardiology, Rigshospitalet

REFERENCES:
- [Derived] Monk-Hansen T, Dall CH, Christensen SB, Snoer M, Gustafsson F, Rasmusen H, Prescott E. Interval training does not modulate diastolic function in heart transplant recipients. Scand Cardiovasc J. 2014 Apr;48(2):91-8. doi: 10.3109/14017431.2013.871058. Epub 2014 Jan 27. PMID 24320690